CLINICAL TRIAL: NCT04363710
Title: Prospective Interventional Study on Reversibility of Type 2 Diabetes Mellitus With Hypocaloric Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Max Healthcare Insititute Limited (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RT2DM20
Record Dates: First submitted 2020-04-13; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Type 2 Diabetes Mellitus in Obese
Keywords: Type 2 Diabetes Mellitus, Low Calorie Diet, Meal Replacer
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in this arm were advised intervention of Low Calorie Diet (800-1000 Kcal/day) for 8 weeks without any anti diabetic medication
  Interventions: Other: Low Calorie Diet
- Control Group (No Intervention): Participants in this arm were kept on their standard medical treatment

INTERVENTIONS:
Other: Low Calorie Diet — 800-1000 Kcal/day
  Arms: Intervention group

SUMMARY:
T2DM, a chronic progressive disorder has an epidemic status in India. Remission (HbA1c of < 6.5% without any anti-diabetic medication) of T2DM is achievable with diet modifications in recently diagnosed obese T2D individuals. Studies suggest Very Low Calorie Diet (600 - 800kcal) and Low Calorie Diet-LCD (800 -1000 kcal) using Meal replacers (MR) are helpful. The investigators aimed to study the effects of LCD without any anti diabetic medication in intervention group and later comparing it with Control group (on standard medical treatment).

DETAILED DESCRIPTION:
The objective is to study the effect of LCD in anthropometric , biochemical and NAFLD (Non Alcholic Fatty Liver Disease) parameters after 8 weeks and 24 weeks from enrollment.

Purposive sampling is used to enroll participants in the study. The LCD is a combination of one meal replacer and modified major meals. Calculated exchanges of food groups is taken care of in the other two major meals and snacks in between. Inorder to adhere compliance clinical (at baseline, after 8 weeks, after 24 weeks) as well as virtual visits through whatsapp, e-mails, SMS, phone calls (once a week during 8 weeks of intervention and further once a month upto 24 weeks) are scheduled. After 8 weeks of LCD, calorie is increased to 1200-1400 Kcal/day. In the control group the standard medical treatment is continued.

The data is collected in case report form and analysed using SPSS software by statistician.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BMI ≥ 30 kg/m^2
* DM history of less than 6 years.
* HBA1C of 6.5-8.5 %.
* On two or less than two diabetes medication.

Exclusion Criteria:

* Patients on Insulin
* Patients having any co morbidity like severe diabetic nephropathy, neuropathy and any other serious illness.
* Evidence of Type 1 diabetes, ketones and acidosis.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
HbA1c in percentage | up to 24 weeks
  To bring HbA1c below diagnostic criteria of type 2 diabetes mellitus as per ADA 2020
Fasting Blood Glucose in millimoles per liter and Fasting Insulin Level in picomole per liter will be combined to report HOMA IR | up to 24 weeks
  To achieve normal HOMA IR range
Weight in kilogram and height in meters will be combined to report BMI in Kg/m^2 | up to 24 weeks
  when obese T2D individuals will have significant improvement in BMI

CONTACTS AND LOCATIONS:
Overall Officials: Sujeet Jha, MRCP, Principal Investigator — Prinicipal Director, Institute of Endocrinology & Metabolism, Maxhealthcare
Locations (1):
- Max Healthcare, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No